CLINICAL TRIAL: NCT03233737
Title: A Double-blind, Cross-over, Incomplete Factorial Study to Assess the Local Anesthetic Efficacy and Safety of CTY-5339 Anesthetic Spray (CTY-5339A) When Applied to the Gingival Mucosal Tissue in Normal Volunteers
Brief Title: Pain Study to Assess Local Anesthetic Efficacy and Safety of CTY-5339 on Gingival Mucosal Tissue in Normal Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cetylite Industries (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: C-003
Record Dates: First submitted 2017-07-26; First posted 2017-07-31 (Actual); Results first posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: No Disease State or Condition
Keywords: local anesthesia; pain tolerance; experimental pain
MeSH Terms: interventions — Benzocaine; Tetracaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Stage II: One spray CTY-5339-A, then one spray CTY-5339-CB (Experimental): A single spray of CTY-5339-A Anesthetic Spray (14.0% benzocaine and 2.0% tetracaine HCl) tested over a 60 minute session, followed by a 4-14 day washout period, followed by a single spray of CTY-5339-CB Anesthetic Spray (14.0% benzocaine) tested over a 60 minute session. Used in Stage II of the study only.
  Interventions: Combination Product: One spray CTY-5339-A; Device: One spray CTY-5339-CB
- Stage II: One spray of CTY-5339-CB, then one spray CTY-5339-A (Active Comparator): A single spray of CTY-5339-CB Anesthetic Spray (14.0% benzocaine) tested over a 60 minute session, followed by a 4-14 day washout period, followed by a single spray of CTY-5339-A Anesthetic Spray (14.0% benzocaine and 2.0% tetracaine HCl) tested over a 60 minute session. Used in Stage II of the study only.
  Interventions: Combination Product: One spray CTY-5339-A; Device: One spray CTY-5339-CB
- Stage I: One spray CTY-5339-A (Experimental): Metered spray bottle with ≈200 uL total spray volume. Contains the active ingredients: 14.0% Benzocaine (USP = 28 mg) and 2.0% Tetracaine Hydrochloride (USP = 4 mg). Administered in a single anesthetic spray. Tested over a 60 minute session. Used in Stage I of the study only.
  Interventions: Combination Product: One spray CTY-5339-A
- Stage I: One spray CTY-5339-CB (Active Comparator): Metered spray bottle with ≈200 uL total spray volume. Contains the active ingredient: 14.0% Benzocaine (USP = 28 mg). Administered in a single anesthetic spray. Tested over a 60 minute session. Used in Stage I of the study only.
  Interventions: Device: One spray CTY-5339-CB
- Stage I: One spray CTY-5339-P (Placebo Comparator): Metered spray bottle with ≈200 uL total spray volume. Contains no active ingredient (placebo: vehicle control). Administered in a single anesthetic spray. Tested over a 60 minute session. Used in Stage I of the study only.
  Interventions: Device: One spray CTY-5339-P

INTERVENTIONS:
Combination Product: One spray CTY-5339-A — Metered spray bottle with ≈200 uL total spray volume. Contains the active ingredients: 14.0% Benzocaine (USP = 28 mg) and 2.0% Tetracaine Hydrochloride (USP = 4 mg). Administered in a single anesthetic spray.
  Other Names: CTY-5339-A; CTY-5339 Anesthetic Spray; benzocaine; tetracaine; tetracaine HCl; 14.0% benzocaine; 2.0% tetracaine HCl; 2.0% tetracaine; 14.0% benzocaine and 2.0% tetracaine HCl; 14.0% benzocaine and 2.0% tetracaine; benzocaine and tetracaine HCl; benzocaine and tetracaine
  Arms: Stage I: One spray CTY-5339-A; Stage II: One spray CTY-5339-A, then one spray CTY-5339-CB; Stage II: One spray of CTY-5339-CB, then one spray CTY-5339-A
Device: One spray CTY-5339-CB — Metered spray bottle with ≈200 uL total spray volume. Contains the active ingredient: 14.0% Benzocaine (USP = 28 mg). Administered in a single anesthetic spray.
  Other Names: CTY-5339-CB; benzocaine; 14.0% benzocaine
  Arms: Stage I: One spray CTY-5339-CB; Stage II: One spray CTY-5339-A, then one spray CTY-5339-CB; Stage II: One spray of CTY-5339-CB, then one spray CTY-5339-A
Device: One spray CTY-5339-P — Placebo. Metered spray bottle with ≈200 uL total spray volume. Contains no active ingredient (vehicle control).
  Other Names: CTY-5339-P; placebo; vehicle control
  Arms: Stage I: One spray CTY-5339-P

SUMMARY:
The purpose of this study is to determine if the topical application to gingival tissue of the combination of benzocaine and tetracaine has a longer duration of local anesthetic activity than benzocaine alone.

DETAILED DESCRIPTION:
In a blinded study, either benzocaine alone or the combination of benzocaine and tetracaine will be sprayed onto the gingival mucosal tissue. Onset and duration of local anesthesia will be evaluated over a one hour period using pin prick and quantitative sensory testing of heat (QST-heat) stimulation. Subjects will receive both treatments in a cross-over design with each session separated by 4-14 days. A total of 50 subjects (normal volunteers) will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between 18-75 years of age with a Body Mass Index (BMI) ≤32;
* Subjects are category I or II on the American Society of Anesthesiologists physical status classification system (ASA category I or II) and are in normal physical health as judged by physical and laboratory examinations;
* Subjects have normal appearance of the oral mucosal tissues;
* At screening and at Baseline during Stage 1 and Sessions 1 and 2, of Stage 2 subjects with Pin-Prick-Test (PPT) scores of at least "3" (on a 10 point numerical rating scale [NRS]) on the 2 readings, 1 of which must be a score of at least "4";
* Subjects have mean quantitative sensory test of heat (QST-Heat) pain sensation temperature assessments on the gingival mucosa of 46.5 °C or less based on the average of the 2 readings at screening and at the Baseline Study Sessions for Stages 1 and 2;
* Subjects must agree to refrain from ingesting any systemic or topical analgesic medication for 3 days or 5 half-lives of the drug prior to and during the study period and alcohol for 1 day prior to and during the study period;
* Subjects must agree to refrain from using mouth rinses, cough drops or throat lozenges on the day of each test session;
* Female subjects must be physically incapable of childbearing potential (postmenopausal for more than 1 year or surgically sterile) or practicing an acceptable method of contraception (hormonal, barrier with spermicide, intrauterine device, vasectomized or same sex partner, or abstinence). Subjects using hormonal birth control must have been on a stable dose of treatment for at least 30 days and received at least 1 cycle of treatment prior to randomization. At Screening and at Baseline of both sessions, all females of childbearing potential must have a negative urine pregnancy test and not be breastfeeding;
* Negative urine drug screen for drugs of abuse at Screening and at Baseline for each Study Session. A positive drug screen result may be permitted if the subject has been on a stable dose of an allowed medication for >30 days;
* Subjects must be capable of reading, comprehending, and signing the informed consent form.

Exclusion Criteria:

* Subjects with a history of any significant hepatic, renal, endocrine, cardiac, neurological, psychiatric, gastrointestinal, pulmonary, hematologic, or metabolic disorders, including glaucoma, diabetes, emphysema, and chronic bronchitis;
* Subjects with a history of any type of cancer other than skin related cancers;
* Subjects with conditions that affect the absorption, metabolism, or passage of drugs out of the body, (e.g., sprue, celiac disease, Crohn's disease, colitis, or liver, kidney, or thyroid conditions);
* Subjects with any history of alcohol or substance abuse (including a positive drug screen test);
* Subjects that currently have or have a history of uncontrolled hypertension;
* Subjects with a known hypersensitivity to any local anesthetic drug;
* Subjects with a hematocrit level significantly below the normal range on the screening laboratory examination (as judged by the PI);
* Subjects with any clinically significant abnormal lab result (as judged by the PI);
* Subjects with any condition or history felt by the Investigator to place the subject at increased risk;
* Subjects who have smoked or chewed tobacco-containing substances within 6 months prior to the start of the study;
* Subjects judged by the Investigator to be unable or unwilling to comply with the requirements of the protocol;
* Subjects who have used an investigational drug within 30 days prior to entering the study;
* Subjects who have donated blood within 3 months prior to the start of the study;
* Subjects who have previously participated in the trial;
* Subjects who are members of the study site staff directly involved with the study or a relative of the Sponsor or other personnel involved with the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen A Cooper, DMD, PhD, Study Chair
Locations (1):
- University of Pennsylvania, School of Dental Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hersh EV, Secreto S, Wang S, Giannakopoulos H, Mousavian M, Lesavoy B, Hutcheson MC, Farrar JT, Wang P, Doyle G, Cooper SA. A Proof-of-concept Study Using Quantitative Sensory Threshold Analysis to Compare Two Intraoral Topical Anesthetics. Clin Ther. 2019 Feb;41(2):291-302. doi: 10.1016/j.clinthera.2018.12.009. Epub 2019 Jan 17. PMID 30660443

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stage I: One Spray CTY-5339-A | Stage I: One Spray CTY-5339-CB | Stage I: One Spray CTY-5339-P | Stage II: One Spray CTY-5339-A, Then One Spray CTY-5339-CB | Stage II: One Spray of CTY-5339-CB, Then One Spray CTY-5339-A
Started | 10 | 10 | 5 | 24 | 26
Completed | 10 | 10 | 5 | 24 | 26
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stage II: One Spray CTY-5339-A, Then One Spray CTY-5339-CB | Stage II: One Spray of CTY-5339-CB, Then One Spray CTY-5339-A | Stage I: One Spray CTY-5339-A | Stage I: One Spray CTY-5339-CB | Stage I: One Spray CTY-5339-P | Total
Number analyzed (Participants) | 24 | 26 | 10 | 10 | 5 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.3 (4.9) | 23.5 (1.8) | 28.1 (6.0) | 27.6 (2.5) | 26.2 (2.4) | 25.1 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 21 | 4 | 8 | 1 | 49
  Male | 9 | 5 | 6 | 2 | 4 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 2 | 1 | 2 | 8
  Not Hispanic or Latino | 24 | 23 | 8 | 9 | 3 | 67
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 8 | 12 | 4 | 5 | 1 | 30
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 0 | 0 | 2
  White | 13 | 12 | 5 | 5 | 3 | 38
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 0 | 0 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 24 | 26 | 10 | 10 | 5 | 75
Weight (lbs) [Mean (Standard Deviation); unit: lbs] | 154.1 (33.0) | 141.2 (27.6) | 151.6 (31.0) | 128.1 (22.5) | 166.0 (35.4) | 146.6 (29.9)
Height (inches) [Mean (Standard Deviation); unit: inches] | 67.3 (4.1) | 65.8 (2.6) | 66.9 (4.2) | 65.1 (1.9) | 67.2 (2.3) | 66.4 (3.3)

OUTCOME MEASURES:

1. Primary Outcome: Stage II: Duration of Anesthesia as Measured by Pin Prick Test (PPT) for One Spray CTY-5339-A Compared to One Spray CTY-5339-CB
Description: The duration of effect, was defined as the length of time in minutes from onset of anesthesia to the absence of anesthesia.Onset was the time point at which the PPT average pain score was less than the Baseline PPT average score by any amount. Also, in 10 minutes or less, the subject must have had a lower PPT average pain score of ≥ 1 unit than Baseline. Absence of anesthesia was defined as follows: After Onset had been established, absence was the first of two time points with consecutive occurrences of regression of absence of analgesia. Reports of less pain by ≥1 unit than Baseline indicated analgesia; while a report of similar (< 1 unit) or more pain than Baseline indicated regression or absence of analgesia. The minimum onset time was 1 minute. PPT scores were assessed using a 0 (no pain) to 10 (severe pain) Numerical Rating Scale at a frequency of every 1 minute for the first 5 minutes and then every 5 minutes thereafter until the final 60 minute time point.
  Stage II outcome.
Time Frame: Up to one hour post-application
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- One Spray CTY-5339-A: Metered spray bottle with ≈200 uL total spray volume. Contains the active ingredients: 14.0% Benzocaine (USP = 28 mg) and 2.0% Tetracaine Hydrochloride (USP = 4 mg). Administered in a single anesthetic spray. Tested over a 60 minute session.
- One Spray CTY-5339-CB: Metered spray bottle with ≈200 uL total spray volume. Contains the active ingredient: 14.0% Benzocaine (USP = 28 mg). Administered in a single anesthetic spray. Tested over a 60 minute session.
Arm/Group | One Spray CTY-5339-A | One Spray CTY-5339-CB
Number analyzed (Participants) | 50 | 50
minutes | 14.6 (16.1) | 7.4 (11.1)

2. Primary Outcome: Stage II: Duration of Anesthesia as Measured by Heat Sensation Threshold (QST Heat) for One Spray CTY-5339-A Compared to One Spray CTY-5339-CB
Description: The duration of effect, was defined as the time from onset to treatment failure, as measured by QST Heat score. QST Heat scores were the temperature where the sensation of a heat stimuli was felt: ranging from 35 ºC to a maximum of 50.5 ºC with intervals of 0.5 ºC, at a frequency of every 1 minute for the first 5 minutes and then every 5 minutes thereafter until the final 60 minute time point. The QST Heat-based "Duration of effect" was calculated by the length of time in minutes from onset of anesthesia to the absence of anesthesia where Onset of anesthesia was defined by PPT unless specific QST thresholds were not met. After Onset had been established, absence of analgesia or offset was the first of two time points with consecutive occurrences of regression or absence of analgesia. Reports of QST heat pain temperature by ≥ 3 °C of the Baseline QST indicated analgesia; while a report of similar (<3 °C) than Baseline indicated regression or absence of analgesia. Stage
Time Frame: Up to one hour post-application
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | One Spray CTY-5339-A | One Spray CTY-5339-CB
Number analyzed (Participants) | 50 | 50
minutes | 45.5 (13.6) | 40.8 (16.3)

3. Primary Outcome: Stage I: Duration of Anesthesia as Measured by Pin Prick Test (PPT) for One Spray CTY-5339-A Compared to One Spray CTY-5339-CB Compared to One Spray CTY-5339-P (Placebo: Vehicle Control)
Description: The duration of effect, was defined as the length of time in minutes from onset of anesthesia to the absence of anesthesia.Onset was the time point at which the PPT average pain score was less than the Baseline PPT average score by any amount. Also, in 10 minutes or less, the subject must have had a lower PPT average pain score of ≥ 1 unit than Baseline. Absence of anesthesia was defined as follows: After Onset had been established, absence was the first of two time points with consecutive occurrences of regression of absence of analgesia. Reports of less pain by ≥1 unit than Baseline indicated analgesia; while a report of similar (< 1 unit) or more pain than Baseline indicated regression or absence of analgesia. The minimum onset time was 1 minute. PPT scores were assessed using a 0 (no pain) to 10 (severe pain) Numerical Rating Scale at a frequency of every 1 minute for the first 5 minutes and then every 5 minutes thereafter until the final 60 minute time point.
  Stage I outcome.
Time Frame: Up to one hour post-application
Population: Placebo duration of effect was not analyzed.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Stage I: One Spray CTY-5339-A | Stage I: One Spray CTY-5339-CB | Stage I: One Spray CTY-5339-P
Number analyzed (Participants) | 10 | 10 | 5
minutes | 49.2 (14.34) | 21.3 (15.47) | 25.2 (30.9)

4. Primary Outcome: Stage I: Duration of Anesthesia as Measured by Heat Sensation Threshold (QST Heat) for One Spray CTY-5339-A Compared to One Spray CTY-5339-CB Compared to One Spray CTY-5339-P (Placebo: Vehicle Control)
Description: The duration of effect, was defined as the time from onset to treatment failure, as measured by QST Heat score. QST Heat scores were the temperature where the sensation of a heat stimuli was felt: ranging from 35 ºC to a maximum of 50.5 ºC with intervals of 0.5 ºC, at a frequency of every 1 minute for the first 5 minutes and then every 5 minutes thereafter until the final 60 minute time point. The QST Heat-based "Duration of effect" was calculated by the length of time in minutes from onset of anesthesia to the absence of anesthesia where Onset of anesthesia was defined by PPT unless specific QST thresholds were not met. After Onset had been established, absence of analgesia or offset was the first of two time points with consecutive occurrences of regression or absence of analgesia. Reports of QST heat pain temperature by ≥ 3 °C of the Baseline QST indicated analgesia; while a report of similar (<3 °C) than Baseline indicated regression or absence of analgesia. Stage I outcome.
Time Frame: Up to one hour post-application
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Stage I: One Spray CTY-5339-A | Stage I: One Spray CTY-5339-CB | Stage I: One Spray CTY-5339-P
Number analyzed (Participants) | 10 | 10 | 5
minutes | 42.5 (21.10) | 6.1 (11.49) | 5 (9.3)

5. Secondary Outcome: Stage II: Onset of Anesthesia for Pin Prick Test (PPT)
Description: Onset of anesthesia was the time point at which the PPT average pain score was less than the Baseline PPT average score by any amount. Also, in 10 minutes or less, the subject must have had a lower PPT average pain score of ≥ 1 unit than the Baseline PPT. Onset was expected to be between 1 and 5 minutes. PPT scores were assessed using a 0 (no pain) to 10 (severe pain) Numerical Rating Scale at a frequency of every 1 minute for the first 5 minutes and then every 5 minutes thereafter until the final 60 minute time point.
  Stage II outcome.
Time Frame: Up to one hour post-application
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | One Spray CTY-5339-A | One Spray CTY-5339-CB
Number analyzed (Participants) | 50 | 50
minutes | 1.1 (0.2) | 1.1 (0.6)

6. Secondary Outcome: Stage II: Onset of Anesthesia for Heat Sensation Threshold (QST Heat)
Description: Onset of anesthesia was defined by Pin Prick Test (PPT) unless specific QST thresholds were not met.
  * If the PPT Onset was 5 minutes or less, then QST must have been greater than the Baseline QST temperature at 5 minutes by any amount and QST must have been ≥ 3 °C of the Baseline QST at 5 or 10 minutes.
  * If the PPT Onset was 10 minutes, then QST must have been ≥ 3 °C of the Baseline QST temperature at 10 minutes.
  * If PPT did not achieve Onset, then QST alone could have achieved onset at either 5 or 10 minutes if QST was greater than the Baseline QST temperature at 5 or 10 minutes by any amount and the QST was ≥ 3 °C of the Baseline QST at 5 or 10 minutes.
  QST Heat scores were the temperature where the sensation of a heat stimuli was felt: ranging from 35 ºC to a maximum of 50.5 ºC with intervals of 0.5 ºC, at a frequency of every 1 minute for the first 5 minutes and then every 5 minutes thereafter until the final 60 minute time point.
  Stage II outcome.
Time Frame: Up to one hour post-application
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | One Spray CTY-5339-A | One Spray CTY-5339-CB
Number analyzed (Participants) | 50 | 50
minutes | 1 (1.4) | 1.3 (2.4)

7. Secondary Outcome: Stage II: Percentage of Responders for Pin Prick Test (PPT) at Each Time Point
Description: Response at at time point is defined as when the PPT average pain score was less than the Baseline PPT average score by any amount. PPT scores were assessed using a 0 (no pain) to 10 (severe pain) Numerical Rating Scale at a frequency of every 1 minute for the first 5 minutes and then every 5 minutes thereafter until the final 60 minute time point.
  Stage II outcome.
Time Frame: Up to one hour post-application
Measure: Count of Participants; unit: Participants
Arm/Group | One Spray CTY-5339-A | One Spray CTY-5339-CB
Number analyzed (Participants) | 50 | 50
Participants
  Responded to treatment at the 1 minute time point | 47 | 46
  Responded to treatment at the 2 minute time point | 50 | 48
  Responded to treatment at the 3 minute time point | 50 | 48
  Responded to treatment at the 4 minute time point | 49 | 48
  Responded to treatment at the 5 minute time point | 49 | 49
  Responded to treatment at the 10 minute time point | 49 | 49
  Responded to treatment at the 15 minute time point | 49 | 48
  Responded to treatment at the 20 minute time point | 49 | 46
  Responded to treatment at the 25 minute time point | 48 | 45
  Responded to treatment at the 30 minute time point | 46 | 42
  Responded to treatment at the 35 minute time point | 43 | 34
  Responded to treatment at the 40 minute time point | 36 | 27
  Responded to treatment at the 45 minute time point | 32 | 21
  Responded to treatment at the 50 minute time point | 25 | 20
  Responded to treatment at the 55 minute time point | 20 | 20
  Responded to treatment at the 60 minute time point | 19 | 18

8. Secondary Outcome: Stage II: Percentage of Responders for Heat Sensation Threshold (QST Heat) at Each Time Point
Description: Response at a time point is defined as an increase of QST heat pain temperature by ≥ 3 degrees C compared to the Baseline QST.
  QST Heat scores were the temperature where the sensation of a heat stimuli was felt: ranging from 35 ºC to a maximum of 50.5 ºC with intervals of 0.5 ºC, at a frequency of every 1 minute for the first 5 minutes and then every 5 minutes thereafter until the final 60 minute time point.
  Stage II outcome.
Time Frame: Up to one hour post-application
Measure: Count of Participants; unit: Participants
Arm/Group | One Spray CTY-5339-A | One Spray CTY-5339-CB
Number analyzed (Participants) | 50 | 50
Participants
  Responded to treatment at the 1 minute time point | 36 | 29
  Responded to treatment at the 2 minute time point | 37 | 30
  Responded to treatment at the 3 minute time point | 37 | 30
  Responded to treatment at the 4 minute time point | 37 | 30
  Responded to treatment at the 5 minute time point | 37 | 31
  Responded to treatment at the 10 minute time point | 38 | 34
  Responded to treatment at the 15 minute time point | 38 | 31
  Responded to treatment at the 20 minute time point | 36 | 29
  Responded to treatment at the 25 minute time point | 32 | 24
  Responded to treatment at the 30 minute time point | 28 | 19
  Responded to treatment at the 35 minute time point | 24 | 15
  Responded to treatment at the 40 minute time point | 22 | 15
  Responded to treatment at the 45 minute time point | 19 | 12
  Responded to treatment at the 50 minute time point | 17 | 12
  Responded to treatment at the 55 minute time point | 14 | 11
  Responded to treatment at the 60 minute time point | 13 | 9

9. Secondary Outcome: Stage II: Percentage of Subjects Reaching Minimal Pain on Pin Prick Test (PPT) (≤2 on Numerical Rating Scale Pain Scale)
Description: Response is defined as a subject having a PPT average pain score of ≤2 recorded at any single time point where PPT was performed. PPT scores were assessed using a 0 (no pain) to 10 (severe pain) Numerical Rating Scale at a frequency of every 1 minute for the first 5 minutes and then every 5 minutes thereafter until the final 60 minute time point.
  Stage II outcome.
Time Frame: Any time within one hour post-application
Measure: Count of Participants; unit: Participants
Arm/Group | One Spray CTY-5339-A | One Spray CTY-5339-CB
Number analyzed (Participants) | 50 | 50
Participants | 50 | 50

10. Secondary Outcome: Stage II: Duration of Minimal Pain for Pin Prick Test (PPT) (≤2 on Numerical Rating Scale Pain Scale)
Description: Response at a time point is defined as having the PPT average pain score of ≤2. PPT scores were assessed using a 0 (no pain) to 10 (severe pain) Numerical Rating Scale at a frequency of every 1 minute for the first 5 minutes and then every 5 minutes thereafter until the final 60 minute time point.
  Stage II outcome.
Time Frame: Up to one hour post-application
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | One Spray CTY-5339-A | One Spray CTY-5339-CB
Number analyzed (Participants) | 50 | 50
minutes | 14.6 (16.1) | 7.4 (11.1)

11. Secondary Outcome: Stage II: Percentage of Subjects Reaching Maximum Heat for Heat Sensation Threshold (QST Heat)
Description: QST Heat scores were the temperature where the sensation of a heat stimuli was felt: ranging from 35 ºC to a maximum of 50.5 ºC with intervals of 0.5 ºC, at a frequency of every 1 minute for the first 5 minutes and then every 5 minutes thereafter until the final 60 minute time point. Reaching maximum heat for QST Heat was defined as subjects reaching the maximum temperature without reporting pain at one or more time points.
  Stage II outcome.
Time Frame: Any time within one hour post-application
Measure: Count of Participants; unit: Participants
Arm/Group | One Spray CTY-5339-A | One Spray CTY-5339-CB
Number analyzed (Participants) | 50 | 50
Participants | 7 | 5

12. Secondary Outcome: Stage II: Sum of Pain Intensity Differences (SPID) for Pin Prick Test (PPT) (Post-hoc)
Description: SPID was calculated as a sum of the delta PPT scores at each time point until the designated time point. The delta PPT score is defined as the change in PPT score from baseline. PPT scores were assessed using a 0 (no pain) to 10 (severe pain) Numerical Rating Scale at a frequency of every 1 minute for the first 5 minutes and then every 5 minutes thereafter until the final 60 minute time point.
  The total possible scale range was from -100 (best) to +100 (worst) for SPID at the 30 minute time point, and from -160 (best) to +160 (worst) for SPID at the 60 minute time point Lower scores signify a better outcome (less sensitive to pain than at baseline = less pain with therapy = therapy was more effective).
  Stage II outcome.
Time Frame: Up to one hour post-application
Measure: Mean (Standard Deviation); unit: score
Arm/Group | One Spray CTY-5339-A | One Spray CTY-5339-CB
Number analyzed (Participants) | 50 | 50
score
  SPID at the 30 minute time point | -85.2 (35.9) | -63.2 (29.38)
  SPID at the 60 minute time point | -122.6 (63.52) | -86.6 (53.15)

13. Secondary Outcome: Stage II: Sum of Temperature Differences (STID) for Heat Sensation Threshold (QST Heat) (Post-hoc)
Description: STID was calculated as a sum of the delta QST Heat scores at each time point until the designated time point. The delta QST Heat score is defined as the change in QST Heat score from baseline. QST Heat scores were the temperature where the sensation of a heat stimuli was felt: ranging from 35 ºC to a maximum of 50.5 ºC with intervals of 0.5 ºC, at a frequency of every 1 minute for the first 5 minutes and then every 5 minutes thereafter until the final 60 minute time point.
  The total possible scale range was from -155 ºC (best) to +155 ºC (worst) for STID at the 30 minute time point, and from -248 ºC (best) to +248 ºC (worst) for SPID at the 60 minute time point Lower scores signify a better outcome (less sensitive to pain than at baseline = less pain with therapy = therapy was more effective).
  Stage II outcome.
Time Frame: Up to one hour post-application
Measure: Mean (Standard Deviation); unit: Degrees Celcius (ºC)
Arm/Group | One Spray CTY-5339-A | One Spray CTY-5339-CB
Number analyzed (Participants) | 50 | 50
Degrees Celcius (ºC)
  STID at the 30 minute time point | 136.5 (67.78) | 96.6 (72.63)
  STID at the 60 minute time point | 214 (140.10) | 149.1 (142.36)

14. Secondary Outcome: Stage I: Percentage of Responders for Pin Prick Test (PPT) at Each Time Point
Description: Response at at time point is defined as when the PPT average pain score was less than the Baseline PPT average score by any amount. PPT scores were assessed using a 0 (no pain) to 10 (severe pain) Numerical Rating Scale at a frequency of every 1 minute for the first 5 minutes and then every 5 minutes thereafter until the final 60 minute time point.
  Stage I outcome.
Time Frame: Time of application up to one hour post-application
Measure: Count of Participants; unit: Participants
Arm/Group | Stage I: One Spray CTY-5339-A | Stage I: One Spray CTY-5339-CB | Stage I: One Spray CTY-5339-P
Number analyzed (Participants) | 10 | 10 | 5
Participants
  Responded to treatment at the 1 minute time point | 8 | 8 | 4
  Responded to treatment at the 2 minute time point | 9 | 10 | 3
  Responded to treatment at the 3 minute time point | 10 | 10 | 3
  Responded to treatment at the 4 minute time point | 10 | 10 | 3
  Responded to treatment at the 5 minute time point | 10 | 10 | 2
  Responded to treatment at the 10 minute time point | 10 | 10 | 3
  Responded to treatment at the 15 minute time point | 10 | 8 | 3
  Responded to treatment at the 20 minute time point | 10 | 4 | 2
  Responded to treatment at the 25 minute time point | 9 | 4 | 2
  Responded to treatment at the 30 minute time point | 9 | 2 | 2
  Responded to treatment at the 35 minute time point | 9 | 2 | 2
  Responded to treatment at the 40 minute time point | 8 | 1 | 2
  Responded to treatment at the 45 minute time point | 7 | 1 | 2
  Responded to treatment at the 50 minute time point | 7 | 1 | 2
  Responded to treatment at the 55 minute time point | 6 | 1 | 2
  Responded to treatment at the 60 minute time point | 6 | 1 | 2

15. Secondary Outcome: Stage I: Percentage of Responders for Heat Sensation Threshold (QST Heat) at Each Time Point
Description: Response at a time point is defined as an increase of QST heat pain temperature by ≥ 3 degrees C compared to the Baseline QST. QST Heat scores were the temperature where the sensation of a heat stimuli was felt: ranging from 35 ºC to a maximum of 50.5 ºC with intervals of 0.5 ºC, at a frequency of every 1 minute for the first 5 minutes and then every 5 minutes thereafter until the final 60 minute time point.
  Stage I outcome.
Time Frame: Time of application up to one hour post-application
Measure: Count of Participants; unit: Participants
Arm/Group | Stage I: One Spray CTY-5339-A | Stage I: One Spray CTY-5339-CB | Stage I: One Spray CTY-5339-P
Number analyzed (Participants) | 10 | 10 | 5
Participants
  Responded to treatment at the 1 minute time point | 7 | 2 | 4
  Responded to treatment at the 2 minute time point | 7 | 3 | 4
  Responded to treatment at the 3 minute time point | 8 | 3 | 4
  Responded to treatment at the 4 minute time point | 8 | 3 | 4
  Responded to treatment at the 5 minute time point | 8 | 3 | 4
  Responded to treatment at the 10 minute time point | 9 | 3 | 4
  Responded to treatment at the 15 minute time point | 9 | 2 | 4
  Responded to treatment at the 20 minute time point | 9 | 2 | 4
  Responded to treatment at the 25 minute time point | 9 | 1 | 1
  Responded to treatment at the 30 minute time point | 8 | 1 | 0
  Responded to treatment at the 35 minute time point | 6 | 1 | 0
  Responded to treatment at the 40 minute time point | 6 | 0 | 0
  Responded to treatment at the 45 minute time point | 6 | 0 | 0
  Responded to treatment at the 50 minute time point | 6 | 0 | 0
  Responded to treatment at the 55 minute time point | 6 | 0 | 0
  Responded to treatment at the 60 minute time point | 6 | 0 | 0

16. Secondary Outcome: Stage I: Duration of Minimal Pain for Pin Prick Test (PPT) (≤2 on Numerical Rating Scale Pain Scale)
Description: Response at a time point is defined as having the PPT average pain score of ≤2. PPT scores were assessed using a 0 (no pain) to 10 (severe pain) Numerical Rating Scale at a frequency of every 1 minute for the first 5 minutes and then every 5 minutes thereafter until the final 60 minute time point.
  Stage I outcome.
Time Frame: Up to one hour post-application
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Stage I: One Spray CTY-5339-A | Stage I: One Spray CTY-5339-CB | Stage I: One Spray CTY-5339-P
Number analyzed (Participants) | 10 | 10 | 5
minutes | 14.5 (11.7) | 2.9 (3.3) | 0.2 (0.4)

17. Secondary Outcome: Stage I: Percentage of Subjects Reaching Maximum Heat for Heat Sensation Threshold (QST Heat)
Description: QST Heat scores were the temperature where the sensation of a heat stimuli was felt: ranging from 35 ºC to a maximum of 50.5 ºC with intervals of 0.5 ºC, at a frequency of every 1 minute for the first 5 minutes and then every 5 minutes thereafter until the final 60 minute time point. Reaching maximum heat for QST Heat was defined as subjects reaching the maximum temperature without reporting pain at one or more time points.
  Stage I outcome.
Time Frame: Any time within one hour post-application
Measure: Count of Participants; unit: Participants
Arm/Group | Stage I: One Spray CTY-5339-A | Stage I: One Spray CTY-5339-CB | Stage I: One Spray CTY-5339-P
Number analyzed (Participants) | 10 | 10 | 5
Participants | 5 | 0 | 0

18. Secondary Outcome: Stage I: Onset of Anesthesia for Pin Prick Test (PPT)
Description: Onset of anesthesia was the time point at which the PPT average pain score was less than the Baseline PPT average score by any amount. Also, in 10 minutes or less, the subject must have had a lower PPT average pain score of ≥ 1 unit than the Baseline PPT. Onset was expected to be between 1 and 5 minutes. PPT scores were assessed using a 0 (no pain) to 10 (severe pain) Numerical Rating Scale at a frequency of every 1 minute for the first 5 minutes and then every 5 minutes thereafter until the final 60 minute time point.
  Stage I outcome.
Time Frame: Up to one hour post-application
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Stage I: One Spray CTY-5339-A | Stage I: One Spray CTY-5339-CB | Stage I: One Spray CTY-5339-P
Number analyzed (Participants) | 10 | 10 | 5
minutes | 1.3 (0.7) | 1.2 (0.4) | 2.8 (4.0)

19. Secondary Outcome: Stage I: Onset of Anesthesia for Heat Sensation Threshold (QST Heat)
Description: Onset of anesthesia was defined by Pin Prick Test (PPT) unless specific QST thresholds were not met.
  * If the PPT Onset was 5 minutes or less, then QST must have been greater than the Baseline QST temperature at 5 minutes by any amount and QST must have been ≥ 3 °C of the Baseline QST at 5 or 10 minutes.
  * If the PPT Onset was 10 minutes, then QST must have been ≥ 3 °C of the Baseline QST temperature at 10 minutes.
  * If PPT did not achieve Onset, then QST alone could have achieved onset at either 5 or 10 minutes if QST was greater than the Baseline QST temperature at 5 or 10 minutes by any amount and the QST was ≥ 3 °C of the Baseline QST at 5 or 10 minutes.
  QST Heat scores were the temperature where the sensation of a heat stimuli was felt: ranging from 35 ºC to a maximum of 50.5 ºC with intervals of 0.5 ºC, at a frequency of every 1 minute for the first 5 minutes and then every 5 minutes thereafter until the final 60 minute time point.
  Stage I outcome.
Time Frame: Up to one hour post-application
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Stage I: One Spray CTY-5339-A | Stage I: One Spray CTY-5339-CB | Stage I: One Spray CTY-5339-P
Number analyzed (Participants) | 10 | 10 | 5
minutes | 2.0 (2.9) | 0.4 (0.7) | 0.8 (0.4)

20. Secondary Outcome: Stage I: Percentage of Subjects Reaching Minimal Pain on Pin Prick Test (PPT) (≤2 on Numerical Rating Scale Pain Scale)
Description: Response is defined as a subject having a PPT average pain score of ≤2 recorded at any single time point where PPT was performed. PPT scores were assessed using a 0 (no pain) to 10 (severe pain) Numerical Rating Scale at a frequency of every 1 minute for the first 5 minutes and then every 5 minutes thereafter until the final 60 minute time point.
  Stage I outcome.
Time Frame: Any time within one hour post-application
Population: Placebo percentage of response was not analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage I: One Spray CTY-5339-A | Stage I: One Spray CTY-5339-CB | Stage I: One Spray CTY-5339-P
Number analyzed (Participants) | 10 | 10 | 5
Participants | 10 | 9 | 2

21. Secondary Outcome: Stage I: Sum of Pain Intensity Differences (SPID) for Pin Prick Test (PPT) (Post-hoc)
Description: SPID was calculated as a sum of the delta PPT scores at each time point until the designated time point. The delta PPT score is defined as the change in PPT score from baseline. PPT scores were assessed using a 0 (no pain) to 10 (severe pain) Numerical Rating Scale at a frequency of every 1 minute for the first 5 minutes and then every 5 minutes thereafter until the final 60 minute time point.
  The total possible scale range was from -100 (best) to +100 (worst) for SPID at the 30 minute time point, and from -160 (best) to +160 (worst) for SPID at the 60 minute time point Lower scores signify a better outcome (less sensitive to pain than at baseline = less pain with therapy = therapy was more effective).
  Stage I outcome.
Time Frame: Up to one hour post-application
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Stage I: One Spray CTY-5339-A | Stage I: One Spray CTY-5339-CB | Stage I: One Spray CTY-5339-P
Number analyzed (Participants) | 10 | 10 | 5
score
  SPID at the 30 minute time point | -82.1 (34.9) | -37.8 (42.3) | -29.3 (36.3)
  SPID at the 60 minute time point | -128.1 (76.6) | -44.0 (52.7) | -53.3 (69.1)

22. Secondary Outcome: Stage I: Sum of Temperature Differences (STID) for Heat Sensation Threshold (QST Heat) (Post-hoc)
Description: STID was calculated as a sum of the delta QST Heat scores at each time point until the designated time point. The delta QST Heat score is defined as the change in QST Heat score from baseline. QST Heat scores were the temperature where the sensation of a heat stimuli was felt: ranging from 35 ºC to a maximum of 50.5 ºC with intervals of 0.5 ºC, at a frequency of every 1 minute for the first 5 minutes and then every 5 minutes thereafter until the final 60 minute time point.
  The total possible scale range was from -155 ºC (best) to +155 ºC (worst) for STID at the 30 minute time point, and from -248 ºC (best) to +248 ºC (worst) for SPID at the 60 minute time point Lower scores signify a better outcome (less sensitive to pain than at baseline = less pain with therapy = therapy was more effective).
  Stage I outcome.
Time Frame: Up to one hour post-application
Measure: Mean (Standard Deviation); unit: Degrees Celcius (ºC)
Arm/Group | Stage I: One Spray CTY-5339-A | Stage I: One Spray CTY-5339-CB | Stage I: One Spray CTY-5339-P
Number analyzed (Participants) | 10 | 10 | 5
Degrees Celcius (ºC)
  STID at the 30 minute time point | 153.0 (72.0) | 10.4 (89.4) | 72.5 (33.6)
  STID at the 60 minute time point | 320.2 (167.2) | 26.1 (137.0) | 134.6 (94.3)

ADVERSE EVENTS:
Time Frame: Adverse event data collected during and for one hour post testing.
Groups:
- One Spray CTY-5339-P: Metered spray bottle with ≈200 uL total spray volume. Contains no active ingredient (placebo: vehicle control). Administered in a single anesthetic spray. Tested over a 60 minute session.
Arm/Group | One Spray CTY-5339-A | One Spray CTY-5339-CB | One Spray CTY-5339-P
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/5
Other Adverse Events (participants affected / at risk) | 2/60 | 2/60 | 0/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | One Spray CTY-5339-A (N=60) | One Spray CTY-5339-CB (N=60) | One Spray CTY-5339-P (N=5)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Mild Headache
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — Mild Nasal Congestion
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — Mild Oropharyngeal pain
Pharyngitis streptococcal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Moderate case of streptococcal pharyngitis
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Mild Pruritus
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Mild Rash

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-24): https://cdn.clinicaltrials.gov/large-docs/37/NCT03233737/Prot_SAP_000.pdf